CLINICAL TRIAL: NCT04798287
Title: Safety of TofAcitinib in Routine Care Patients With Rheumatoid Arthritis (STAR-RA)-Cancer Endpoints
Acronym: STAR-RA-Cancer
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Seoyoung C. Kim, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2011P002580-207
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Tumor Necrosis Factor Inhibitors; Infliximab; Adalimumab; Certolizumab Pegol; Etanercept; golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with Tofacitinib: Real-World Evidence (RWE) and RCT-Duplicate
  Interventions: Drug: Tofacitinib
- Patients treated with TNF inhibitors: Real-World Evidence (RWE) and RCT-Duplicate
  Interventions: Drug: TNF Inhibitor

INTERVENTIONS:
Drug: Tofacitinib — First eligible prescription for treating rheumatoid arthritis (RA)
  Groups: Patients treated with Tofacitinib
Drug: TNF Inhibitor — First eligible prescription for treating rheumatoid arthritis (RA)
  Other Names: infliximab; adalimumab; certolizumab pegol; etanercept; golimumab
  Groups: Patients treated with TNF inhibitors

SUMMARY:
There are two main aims of this study.

First aim is to compare the risk of composite cancer outcomes, between patients treated with tofacitinib and patients treated with TNF inhibitors (TNFi) for rheumatoid arthritis (RA) among, 1) "real world evidence (RWE)" cohorts including routine care patient population from the US and, 2) "Randomized controlled trial (RCT) DUPLICATE" cohorts including routine care patient population who meet inclusion and exclusion criteria of the Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis ("ORAL Surveillance", NCT02092467) clinical trial.

Second aim is to examine the risk of common solid cancers (lung, colorectal, breast, prostate), hematological cancers, and non-melanoma skin cancer as separated endpoints when comparing tofacitinib with TNFi in patients with RA among, 1) "real world evidence (RWE)" cohort including routine care patient population from the US and, 2) "Randomized controlled trial (RCT) DUPLICATE" cohort including routine care patient population who meet inclusion and exclusion criteria of the Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis ("ORAL Surveillance", NCT02092467) clinical trial.

ELIGIBILITY:
Criteria:

Please see https://www.bwhprime.org/resources.html for full code and algorithm definitions.

Eligible cohort entry dates:

* For US MarketScan, 2012-2018
* For Optum, 2012-2020
* For Medicare Claims Database (Parts A, B and D), 2012-2017

Cohort entry date:

* First TNFi or tofacitinib dispensation/administration date

Inclusion and Exclusion Criteria Common to RWE and RCT-duplicate Cohorts:

1. Inclusion Criteria

   * Patients treated with tofacitinib or TNF inhibitors in IBM MarketScan, Optum, and Medicare fee-for-service
   * A minimum of 365 days of continuous enrollment in health plan prior to (and including) the cohort entry date
   * Two diagnosis codes for RA in any setting in 365 days baseline period (diagnosis codes between 7 and 365 days apart)
2. Exclusion Criteria

   * Index drug in 365 days prior to cohort entry date (prevalent users)
   * Missing data on age or gender
   * Admission to nursing facility or hospice on or prior to cohort entry date (ever look-back)
   * Diagnosis of malignant cancer prior to cohort entry date (ever look-back period)
   * TNFi users with history of any Janus kinase (JAK) inhibitors (tofacitinib, upadacitinib, or baricitinib) (ever look-back period)
   * TNFi users initiating with more than one TNFi on same date
   * Tofacitinib users with a prescription of baricitinib, upadacitinib (ever look-back period)
   * Tofacitinib users initiating treatment on multiple JAK inhibitors on same day (tofacitinib and baricitinib, tofacitinib and upadacitinib)

Exclusion criteria specific to RWE cohorts:

* Patients less than 18 years of age (MarketScan and Optum) and 65 years of age (Medicare) at cohort entry

Inclusion criteria specific to RCT-duplicate cohorts:

* Patients with at least one methotrexate dispensation (six months look-back period)
* Patients with at least one cardiovascular risk factor (including smoking, hypertension, dyslipidemia, diabetes mellitus, ischemic heart disease, family history of ischemic heart disease) (one-year look-back period)

Exclusion criteria specific to RCT-duplicate cohorts:

* Patients less than 50 years of age (MarketScan and Optum) and 65 years
* Patients recently hospitalized with infections (30-day look-back period)
* Pregnant patients (one year look-back period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be two independent study populations:
  1. Real-World Evidence (RWE) cohorts: This study population will reflect the patients diagnosed with RA who are routinely treated and managed in setting of clinical practice.
  2. RCT-duplicate cohorts: This study population will emulate "the Safety Study Of Tofacitinib Versus Tumor Necrosis Factor (TNF) Inhibitor In Subjects With Rheumatoid Arthritis" clinical trial ("ORAL Surveillance", NCT02092467). The inclusion and exclusion criteria of this RCT will be applied to this study population.
Sampling Method: Non-Probability Sample
Enrollment: 105711 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Time to second outpatient or inpatient diagnosis of any cancer (excluding NMSC and any carcinoma in situ diagnosis) | Through study time period (2012-2020)

SECONDARY OUTCOMES:
Time to second outpatient or inpatient diagnosis of lung cancer (excluding any carcinoma in situ diagnosis) | Through study time period (2012-2020)
Time to second outpatient or inpatient diagnosis of colorectal cancer (excluding any carcinoma in situ diagnosis) | Through study time period (2012-2020)
Time to second outpatient or inpatient diagnosis of breast cancer (excluding any carcinoma in situ diagnosis) | Through study time period (2012-2020)
Time to second outpatient or inpatient diagnosis of prostate cancer (excluding any carcinoma in situ diagnosis) | Through study time period (2012-2020)
Time to second outpatient or inpatient diagnosis of lymphatic/hematopoietic tissue cancers | Through study time period (2012-2020)
Time to second outpatient or inpatient diagnosis of lymphoma | Through study time period (2012-2020)
Time to second outpatient or inpatient diagnosis of leukemia | Through study time period (2012-2020)
Time to first procedure code occurring within 60 days of an outpatient or inpatient diagnosis of NMSC | Through study time period (2012-2020)

CONTACTS AND LOCATIONS:
Overall Officials: Seoyoung C Kim, MD, ScD, MSCE, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Khosrow-Khavar F, Desai RJ, Lee H, Lee SB, Kim SC. Tofacitinib and Risk of Malignancy: Results From the Safety of Tofacitinib in Routine Care Patients With Rheumatoid Arthritis (STAR-RA) Study. Arthritis Rheumatol. 2022 Oct;74(10):1648-1659. doi: 10.1002/art.42250. Epub 2022 Sep 1. PMID 35643956

DOCUMENTS (1):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04798287/Prot_002.pdf